CLINICAL TRIAL: NCT07169058
Title: The Effect of Fascial Mobilization Along the Course of the Vagus Nerve on Acute Physiological Parameters in Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Fascial Mobilization Along the Vagus Nerve and Its Effects on Acute Physiological Parameters in Obstructive Sleep Apnea
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Engin Ramazanoglu, Assistant Professor, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/2-11
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea Syndromes
Keywords: Sleep Apnea, Obstructive; Vagus Nerve; Autonomic Nervous System; Fascial Mobilization
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized controlled trial with two parallel groups. Participants diagnosed with moderate to severe obstructive sleep apnea syndrome will be randomly assigned to either the fascial mobilization group or the control group. The intervention group will receive 16 minutes of manual fascial mobilization along anatomical regions associated with the vagus nerve, while the control group will rest in a supine position for the same duration. The study aims to evaluate acute physiological responses including heart rate, systolic and diastolic blood pressure, and oxygen saturation before and after the intervention.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation. Physiotherapists performing the mobilization were not involved in the measurement process. A different physiotherapist, who was unaware of the participants' group assignments, recorded heart rate, blood pressure, and oxygen saturation before and after the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus Nerve Fascial Mobilization (Experimental): Participants in this group will receive manual fascial mobilization along anatomical regions associated with the vagus nerve, including the occipitomastoid suture, anterior and posterior cervical regions, hyoid, sternum, diaphragm, Trigonum Labbe, and radix mesenteri. Mobilization will be applied for a total of 16 minutes using gentle manual pressure and stretching techniques by a physiotherapist. Heart rate, systolic and diastolic blood pressure, and oxygen saturation will be measured before and after the intervention.
  Interventions: Behavioral: Vagus Nerve Fascial Mobilization
- Sham Control Group (Sham Comparator): Participants in this group will receive a sham procedure. The physiotherapist will place hands on the same anatomical regions for 16 minutes without applying mobilization or therapeutic pressure. No active fascial mobilization will be performed. Heart rate, systolic and diastolic blood pressure, and oxygen saturation will be recorded before and after the sham procedure.
  Interventions: Behavioral: Vagus Nerve Fascial Mobilization

INTERVENTIONS:
Behavioral: Vagus Nerve Fascial Mobilization — Reference Points of the Body Regions for Mobilization
  1. Occipito-Mastoid Suture (OM) The occipitomastoid suture is the cranial suture located between the occipital bone and the mastoid part of the temporal bone. The condylus squamosa mastoidea serves as the pivot point. The patient lies in the supine position while the physiotherapist sits at the head of the patient. One hand is placed under the occiput at the suture, while the other hand is placed on the mastoid portion of the temporal bone. The patient's head is turned toward the direction of mobilization, and mobilization is performed using the weight of the head (25). Each application is planned as a single repetition lasting 120 seconds.
  2. Anterior Cervical Region (Triangle) Topographically, this region is located at the anterior part of the neck, extending along the seven cervical vertebrae (C1-C7). The anterior triangle is bordered superiorly by the lower margin of the mandible, laterally by the anterior median line of the s
  Other Names: 1

SUMMARY:
This randomized controlled trial was designed to investigate the effects of fascial mobilization along the course of the vagus nerve on acute physiological parameters in individuals with obstructive sleep apnea syndrome (OSAS). Patients diagnosed with moderate to severe OSAS by polysomnography at Mardin Training and Research Hospital Sleep Laboratory will be included in the study. Participants will be randomly assigned to mobilization or control groups. In the mobilization group, 16 minutes of manual fascial mobilization will be applied to fascial regions associated with the vagus nerve, starting from the occipitomastoid suture and extending through the cervical, thoracic, and abdominal regions. The control group will rest in the supine position for the same duration. Heart rate, systolic and diastolic blood pressure, and peripheral oxygen saturation (SpO₂) will be recorded before and after the intervention. This study is expected to demonstrate the effectiveness of fascial mobilization as a non-invasive, low-cost, and innovative approach in the treatment of OSAS, contributing to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with moderate to severe obstructive sleep apnea syndrome (OSAS) confirmed by polysomnography (PSG) according to international criteria (AASM - American Academy of Sleep Medicine) with an apnea-hypopnea index (AHI ≥15/hour).

Patients aged between 18 and 65 years.

Patients able to comply with PSG procedures and the manual mobilization protocol.

Patients with stable cardiac and respiratory status.

Patients without acute exacerbations or decompensated disease.

Patients who have not received CPAP, BiPAP, oral appliance therapy, or surgical treatment previously, or who discontinued such treatments at least 3 months prior to enrollment.

Patients not taking medications that directly affect sleep patterns or autonomic nervous system function (e.g., sedatives, hypnotics, anticholinergics).

Patients who provide written informed consent to participate in the study.

Exclusion Criteria:

* Patients with uncontrolled hypertension.

Patients with advanced heart failure, severe arrhythmia, or asthma.

Patients with coronary artery disease.

Patients with a history of cerebrovascular disease.

Patients with chronic obstructive pulmonary disease (COPD).

Patients with interstitial lung disease.

Patients with epilepsy, Parkinson's disease, or dementia.

Patients with major depressive disorder or anxiety disorder.

Patients with a body mass index (BMI) > 40 kg/m².

Patients with a history of major surgery in the cervical region (e.g., thyroidectomy, cervical disc surgery) or vagus nerve injury.

Patients with acute infection, skin lesions, or inflammatory disease in the neck/thoracic region.

Patients currently using CPAP, BiPAP, or oral appliances.

Patients with narcolepsy, insomnia, or parasomnia.

Patients with alcohol use or taking sedative/hypnotic medications.

Patients with night-shift work schedules or irregular sleep patterns.

Pregnant or breastfeeding women.

Patients with cognitive impairment preventing adherence to the study protocol.

Patients with severe musculoskeletal limitations (e.g., in the cervical/thoracic region) that would prevent mobilization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure (mmHg) | Baseline (pre-intervention), immediately post-intervention, 5 minutes post-intervention, and 15 minutes post-intervention.
  Systolic blood pressure will be measured non-invasively using a bedside patient monitor. The outcome will assess changes in systolic blood pressure (mmHg) across time points to evaluate the acute effects of fascial mobilization along the vagus nerve compared with sham procedure.
Heart Rate (beats per minute) | Baseline (pre-intervention), immediately post-intervention, 5 minutes post-intervention, and 15 minutes post-intervention.
  Heart rate will be measured using a bedside patient monitor. The outcome will assess the change in beats per minute (bpm) from baseline (before intervention) to post-intervention. The measure will determine the acute effect of fascial mobilization along the vagus nerve compared with sham procedure.
Diastolic Blood Pressure (mmHg) | Baseline (pre-intervention), immediately post-intervention, 5 minutes post-intervention, and 15 minutes post-intervention.
  Diastolic blood pressure will be measured non-invasively using a bedside patient monitor. The outcome will assess changes in diastolic blood pressure (mmHg) across time points to evaluate the acute effects of fascial mobilization along the vagus nerve compared with sham procedure.
Peripheral Oxygen Saturation (SpO₂, %) | Baseline (pre-intervention), immediately post-intervention, 5 minutes post-intervention, and 15 minutes post-intervention.
  "Peripheral oxygen saturation will be measured using pulse oximetry integrated into the bedside patient monitor. The outcome will assess changes in SpO₂ (%) across time points to evaluate the acute effects of fascial mobilization along the vagus nerve compared with sham procedure."

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Artuklu University, Mardin, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision will depend on journal requirements and ethical committee approval

REFERENCES:
- [Background] Delaney JP, Leong KS, Watkins A, Brodie D. The short-term effects of myofascial trigger point massage therapy on cardiac autonomic tone in healthy subjects. J Adv Nurs. 2002 Feb;37(4):364-71. doi: 10.1046/j.1365-2648.2002.02103.x. PMID 11872106
- [Background] Austelle CW, Cox SS, Wills KE, Badran BW. Vagus nerve stimulation (VNS): recent advances and future directions. Clin Auton Res. 2024 Dec;34(6):529-547. doi: 10.1007/s10286-024-01065-w. Epub 2024 Oct 4. PMID 39363044